CLINICAL TRIAL: NCT04078282
Title: The Use of Collaborative Care in General Practice for Elderly Patients With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Erik L Werner, Professor, University of Oslo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCKO001
Record Dates: First submitted 2019-08-27; First posted 2019-09-06 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Depression in Old Age
Keywords: Depression; Elderly; Family Practice
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial where family physicians are to be randomized into interventional or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment group (Experimental): Patients will meet in a joint consultation with their family physician and a psychiatrist for evaluation. Then it follows three treatment sessions with the family physician before a new joint consultation with the psychiatrist. The intervention ends with three more treatment sessions with the family physician.
  Interventions: Behavioral: Intervention group
- Control group (Active Comparator): Patients belonging to family physicians who constitute the control group will be assessed and given treatment according to usual care. This may include treatment by the family physician, medication, referrals to specialized care.
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Intervention group — see above

SUMMARY:
The first part of this study aims to identify the occurence of depression in the elderly. In the second part, older patients with depression will be invited to a collaborative care with his or her family physician and a psychiatrist specialized in psychiatry in the elderly in accordance with a study protocol. The intervention includes two sessions where the patient will meet the psychiatrist together with the family physician, and between the two sessions the patient will have three treatment sessions with the family physician based on the evaluation by the psychiatrist. Following the last session with the psychiatrist the intervention ends with three more treatment sessions with the family physician.

DETAILED DESCRIPTION:
The frequency of depression in the elderly is little known and experiences from family practice indicate that older people not always communicate their mental health issues or present physical complaints which may arise from a state of depression. In this study we aim to register the occurence of depression among all patients at the age of 65 or older who visit their family physician. During a period of four weeks, all patients meeting the eligibility criteria will be asked to answer a questionnaire about mental and physic health issues. Those who respond in a manner that gives reasons to believe there is a depression will be contacted by their family physician to meet for a consultation and examination. If this examination confirms the diagnosis the patient will either be treated as usual by their family physician (control group) or be invited to a collaborative care with the family physician in cooperation with a psychiatrist who is specialized in psychiatry in the elderly (intervention group). In the control group the patients will receive usual care at their family physician or be referred to a psychiatrist or a psychologist if appropriate. In the intervention group the patients will have a evaluation session with the family physician and the psychiatrist together. Following this session, the patient and the family physician will meet for three treatment consultations based on the evaluation and recommendations given by the psychiatrist. Then there will be one more joint session with the patient, the family physician and the psychiatrist and the whole treatment program ends with three more treatment consultations at the family physician. - The aim of this intervention is to examine whether this treatment program is more or equally efficient to treat depression in the elderly as usual care and at lower cost and use of specialized care.

ELIGIBILITY:
Inclusion Criteria:

* all patients visiting one of the collaborative family physicians during the enrollment period of four weeks

Exclusion Criteria:

* cognitive dysfunction
* speaking Norwegian language

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with a change in clinical significant depression | At start and at 12 and 18 month following treatment
  Change in depression as described by the Patient Health Questionnaire (PHQ-9). The questionnaire is a 9-item questionnaire, each with a 0-4 point scale. A change of 3,9 points in the sumscale is regarded significant.

SECONDARY OUTCOMES:
Number of patients with a change in the level of anxiety | At start and at 12 and 18 month following treatment
  Change in anxiety as described by the Generalized Anxiety Disorder 7-item score GAD-7. The questionnaire is a 7-item questionnaire, each with a 0-4 point scale. There is no consensus on which level of change is regarded significant.
Number of Subjective Health Complaints among patients with depression | At start and at 12 and 18 month following treatment
  Change in subjective Health Complaints as described by the Subjective Health Complaints questionnaire. The questionnaire is a 9-item questionnaire, each with a 0-4 point scale. A change of 3,9 points in the sumscale is regarded significant. The questionnaire is a 29-item questionnaire, each with a 0-4 point scale. There is no consensus on which level of change is regarded significant.

CONTACTS AND LOCATIONS:
Overall Officials: Jørund Straand, PhD, Study Director — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kvalbein-Olsen LC, Aakhus E, Haavet OR, Mdala I, Werner EL. Joint consultations in a structured GP-patient-geriatric-psychiatrist model for late-life depression: a cluster RCT. BMC Prim Care. 2025 Sep 29;26(1):297. doi: 10.1186/s12875-025-03002-w. PMID 41023858